CLINICAL TRIAL: NCT04106297
Title: A First-in-human, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GLPG3970 Single and Multiple Ascending Doses in Adult Healthy Male Subjects, and in Psoriasis Subjects When Administered Daily for 6 Weeks
Brief Title: A Study to Evaluate the Effects of Single and Multiple Oral Doses of GLPG3970
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: GLPG3970-CL-101; 2019-001803-19 (EudraCT Number)
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2021-06

CONDITIONS: Healthy; Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Intervention Model Description: Part 1 and 1bis (SAD), Part 2 (MAD) and Part 4 (psoriasis subjects) are randomized, double-blind, placebo-controlled; Part 3 (FE-rBA) and Part 3bis (FE) are randomized, open-label.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- GLPG3970 SAD (Experimental): Single doses of GLPG3970 at up to 6 dose levels in ascending order
  Interventions: Drug: GLPG3970 oral solution
- Placebo SAD (Placebo Comparator): Single doses of placebo
  Interventions: Drug: Placebo oral solution
- GLPG3970 MAD (Experimental): Multiple doses of GLPG3970 at up to 4 dose levels in ascending order, daily for 14 days
  Interventions: Drug: GLPG3970 oral solution
- Placebo MAD (Placebo Comparator): Multiple doses of placebo
  Interventions: Drug: Placebo oral solution
- GLPG3970 FE-rBA (Experimental): Single dose of GLPG3970 in fed and fasted state
  Interventions: Drug: GLPG3970 oral solution; Drug: GLPG3970 capsule
- GLPG3970 FE (Experimental): Single dose of GLPG3970 in fed and fasted state
  Interventions: Drug: GLPG3970 oral solution
- GLPG3970 in psoriasis subjects (Experimental)
  Interventions: Drug: GLPG3970 oral solution
- Placebo in psoriasis subjects (Experimental)
  Interventions: Drug: Placebo oral solution

INTERVENTIONS:
Drug: GLPG3970 oral solution — GLPG3970 for oral administration
  Arms: GLPG3970 FE; GLPG3970 FE-rBA; GLPG3970 MAD; GLPG3970 SAD; GLPG3970 in psoriasis subjects
Drug: Placebo oral solution — Placebo for oral administration
  Arms: Placebo MAD; Placebo SAD; Placebo in psoriasis subjects
Drug: GLPG3970 capsule — GLPG3970 for oral administration
  Arms: GLPG3970 FE-rBA

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of GLPG3970 in healthy volunteers after single oral administrations of GLPG3970 (SAD), compared to placebo (part 1 and 1bis) and after multiple (for 14 days) oral administrations of GLPG3970 (MAD), compared to placebo (part 2). The effect of food (FE) (high-fat, high calorie) on the pharmacokinetics of GLPG3970 and the relative bioavailability (rBA) of an oral solution versus a solid formulation will be assessed (part 3 and 3bis). Part 4 of the study is to evaluate the safety and tolerability of GLPG3970 in subjects with moderate to severe psoriasis when administered daily for 6 weeks.

ELIGIBILITY:
Inclusion Criteria for Part 1, 1bis, 2, 3 and 3bis:

* Male between 18-55 years of age (extremes included), on the date of signing the informed consent form (ICF).
* A body mass index (BMI) between 18-30 kg/m2, inclusive.
* Judged to be in good health by the investigator based upon the results of a medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), and fasting clinical laboratory safety tests available at screening and prior to randomization. Hemoglobin must not be below the lower limit of normal range. Bilirubin, aspartate aminotransferase (AST), and alanine aminotransferase (ALT) must be no greater than 1.5x upper limit of normal range (ULN). Other clinical laboratory safety test results must be within the reference ranges, or test results that are outside the reference ranges need to be considered not clinically significant in the opinion of the investigator.

This list only contains the key inclusion criteria for the healthy volunteers part of the study.

Inclusion criteria for Part 4:

* Male or female between 18-65 years of age (extremes included), on the date of signing the ICF.
* Diagnosed with plaque psoriasis ≥6 months.
* Screening Psoriasis Area and Severity Index (PASI) ≥12 (moderate to severe) and affected body surface area (BSA) ≥10%.
* A body mass index (BMI) between 18-35 kg/m2, inclusive.

This list only contains the key inclusion criteria for Part 4 of the study.

Exclusion Criteria for Part 1, 1bis, 2, 3 and 3bis:

* Known hypersensitivity to the Investigational Medicinal Product (IMP) ingredients or history of a significant allergic reaction to IMP ingredients as determined by the investigator.
* Positive serology for hepatitis B virus surface antigen (HBsAg) or hepatitis C virus or history of hepatitis from any cause with the exception of hepatitis A that was resolved at least 3 months prior to first dosing of the IMP.
* History of or a current immunosuppressive condition (e.g. human immunodeficiency virus [HIV] infection).

This list only contains the key exclusion criteria for the healthy volunteers part of the study.

Exclusion criteria for Part 4:

* Subject has evidence of skin conditions other than psoriasis (e.g., eczema) at the time of screening or baseline visit that would interfere with the evaluation of psoriasis.
* Subject is unable to discontinue systemic therapies and/or topical therapies for the treatment of psoriasis and cannot discontinue phototherapy (UVB or PUVA) from signing of the ICF up to the end of the study.

This list only contains the key inclusion criteria for Part 4 of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-03-05 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs), treatment-emergent serious adverse events, and TEAEs leading to treatment discontinuations | From screening through study completion, an average of 20 months
  To evaluate the safety and tolerability of GLPG3970 compared to placebo in adult healthy male subjects as single and multiple ascending oral doses, and in subjects with moderate to severe psoriasis when administered daily for 6 weeks

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of GLPG3970 (Part 1 and 1bis) | Between Day 1 pre-dose and Day 4
  To evaluate the pharmacokinetics (PK) of oral SAD of GLPG3970 in adult healthy male subjects
Maximum observed plasma concentration (Cmax) of GLPG3970 (Part 2) | Between Day 1 pre-dose and Day 17
  To evaluate the PK of oral MAD of GLPG3970 in adult healthy male subjects
Maximum observed plasma concentration (Cmax) of GLPG3970 (Part 3 and 3bis, FE) | Between Day 1 pre-dose and Day 4
  To evaluate the food effect on the PK of a single oral dose of GLPG3970 in adult, healthy, subjects
Maximum observed plasma concentration (Cmax) of GLPG3970 (Part 3, rBA) | Between Day 1 pre-dose and Day 4
  To evaluate the PK of a single oral dose of GLPG3970 administered as an oral solution versus and oral capsule in adult, healthy, subjects
Area under curve (AUC) of GLPG3970 (Part 1 and 1bis) | Between Day 1 pre-dose and Day 4
  To evaluate the PK of oral SAD of GLPG3970 in adult healthy male subjects
Area under curve (AUC) of GLPG3970 (Part 2) | Between Day 1 pre-dose and Day 17
  To evaluate the PK of oral MAD of GLPG3970 in adult healthy male subjects
Area under curve (AUC) of GLPG3970 (Part 3 and 3bis, FE) | Between Day 1 pre-dose and Day 4
  To evaluate the food effect on the PK of a single oral dose of GLPG3970 under fed conditions (high-fat high calorie) versus fasted conditions in adult, healthy, subjects
Area under curve (AUC) of GLPG3970 (Part 3, rBA) | Between Day 1 pre-dose and Day 4
  To evaluate the rBA of an oral solution of GLPG3970 versus an oral capsule of GLPG3970 on the PK of a single oral dose of GLPG3970 in adult, healthy, subjects
Terminal elimination half-life (t1/2) of GLPG3970 (Part 1 and 1bis) | Between Day 1 pre-dose and Day 4
  To evaluate the PK of oral SAD of GLPG3970, in adult, healthy, subjects
Terminal elimination half-life (t1/2) of GLPG3970 (Part 2) | Between Day 1 pre-dose and Day 17
  To evaluate the PK of oral MAD of GLPG3970, in adult, healthy, subjects

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Petkova, MD, Study Director — Galapagos NV
Locations (3):
- SGS Belgium NV - Clinical Pharmacology Unit Antwerp, Antwerp, Belgium
- Clinical Republican Hospital Arensia Experimental Medicine, Chisinau, Moldova
- ARENSIA Exploratory Medicine Unit, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No